CLINICAL TRIAL: NCT01023789
Title: ABSORB EXTEND Clinical Investigation: A Continuation in the Clinical Evaluation of the ABSORB Bioresorbable Vascular Scaffold (BVS) System in the Treatment of Subjects With de Novo Native Coronary Artery Lesions
Brief Title: ABSORB EXTEND Clinical Investigation
Acronym: ABSORB EXTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-386; ACTRN12610000131055 (Registry Identifier: Australian New Zealand Clinical Trials Registry); REFCTRI000460, 03-05-2010 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2017-12

CONDITIONS: Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Cardiovascular Disease
Keywords: Drug eluting stent; Stents; Angioplasty; Bioabsorbable; Bioresorbable; Scaffold
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABSORB BVS (Experimental): Absorb Bioresorbable Vascular Scaffold (BVS) System implantation in the treatment of coronary artery disease
  Interventions: Device: ABSORB BVS

INTERVENTIONS:
Device: ABSORB BVS — Absorb Bioresorbable Vascular Scaffold (BVS) System implantation

SUMMARY:
The ABSORB EXTEND trial is to continue the assessment of the safety and performance of the ABSORB Bioresorbable Vascular Scaffold (BVS) System

ABSORB BVS is currently in development at Abbott Vascular.

ELIGIBILITY:
Inclusion Criteria:

* Up to two de novo lesions can be treated, each located in a separate native epicardial vessel.
* Target lesion(s) must be located in a native coronary artery where target vessel(s) diameter is ≥ 2.0 mm and ≤ 3.3 mm and target lesion length is ≤ 28 mm, both assessed by on-line Quantitative Coronary Analysis (QCA).
* Target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1.
* If two treatable lesions meet the inclusion criteria they must be in separate major epicardial vessels (LAD with septal and diagonal branches, left circumflex artery (LCX) with obtuse marginal and/or ramus intermedius branches and right coronary artery (RCA) and any of its branches).
* Percutaneous interventions for lesions in a non-target vessel are allowed if done ≥ 30 days prior to or if planned to be done 6 months after the index procedure.
* Percutaneous intervention for lesions in the target vessel are allowed if done > 6 months prior to or if planned to be done 6 months after the index procedure.

Exclusion Criteria:

* Lesion(s) located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft.
* Lesion(s) involving a bifurcation with side branch vessel ≥ 2 mm in diameter and/or ostial lesion > 40% stenosed by visual estimation or side branch requiring predilatation.
* Total occlusion (TIMI flow 0), prior to wire passing.
* Target vessel(s) contains visible thrombus.
* Another clinically significant lesion is located in the same epicardial vessel (including side branch) as the target lesion(s).
* Subject has received brachytherapy in any epicardial vessel (including side branches).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2010-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Instituto de Cardiologia Dante Pazzanese Unidadae II Recepcao de Angioplastia; Patrick Serruys, MD, Study Chair — Thoraxcenter-Erasmus University
Locations (56):
- Instituto Cardiovascular de Buenos Aires-ICBA, Buenos Aires, Argentina
- Australia (4):
  - Eastern Heart Clinic, The Prince of Wales Hospital, Randwick, New South Wales
  - Wesley Hospital, Auchenflower, Queensland
  - St. Vincent's Hospital, Melbourne, Victoria
  - Monash Medical Center, Melbourne, Victoria
- Allgemeines Krankenhaus Linz, Linz, Austria
- Onze-Lieve VrouweZiekenhuis, Aalst, Belgium
- Brazil (3):
  - Instituto de Cardiologia Dante Pazzanese Unidadae II Recepcao de Angioplastia, São Paulo
  - Sociedade Beneficente Isreaelita Brasileira Hospital Albert Einstein, São Paulo
  - Instituto Coração Triângulo Mineiro, Uberlândia
- Canada (4):
  - Montreal Heart Institute, Montreal
  - University of Ottawa Heart Institute, Ottawa
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
  - St. Michael's Hospital, Toronto
- China (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Århus University Hospital, Århus N, Denmark
- France (3):
  - Institut Jacques Cartier (ICPS), Massy
  - Clinique Pasteur, Toulouse
  - Hopital De Rangueil - CHU, Toulouse
- Germany (2):
  - Charité Berlin Campus Steglitz, Berlin
  - Uni.Klinikum Heidelberg, Heidelberg
- India (8):
  - Apollo Hospital, Hyderabaad, Andhar Pradesh
  - CARE Hospital, Hyderabaad, Andhra Pradesh
  - SAL Hospital And Medical Institute, Ahmedabad
  - Care Institute of Medical Sciences, Ahmedabad
  - Madras Medical Mission, Chennai
  - Medanta -The Medicity, Gūrgaon
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Escorts Heart Institute & Research Centre, New Delhi
- Rabin Medical Center, Petah Tikva, Israel
- Italy (2):
  - Catanzaro University Hospital, Catanzaro
  - Centro Cardiologico Monzino, Milan
- Japan (5):
  - Teikyo University, Tokyo, Itabashi
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Saiseikai Yokohama City Eastern Hospital, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kansai
  - Mitsui Memorial Hospital, Chiyoda-ku
- Institute Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (3):
  - Catharina ZH Eindhoven, Eindhoven
  - Erasmus Medical Center, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
- New Zealand (2):
  - Mercy Angiography Unit, Auckland
  - Christchurch Hospital, Christchurch
- University Hospital Krakow, Krakow, Poland
- National University Hospital, Singapore, Singapore
- Sunninghill Hospital, Johannesburg, South Africa
- Spain (3):
  - Clinico San Carlos, Madrid
  - La Paz, Madrid
  - Hospital do Meixoeiro, Pontevedra
- Lund University Hospital, Lund, Sweden
- Inselspital Bern, Kardiologie, Bern, Switzerland
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - Glenfield Hospital, Leicester
  - King's College Hospital, London

REFERENCES:
- [Derived] Costa JR Jr, Abizaid A, Whitbourn R, Serruys PW, Jepson N, Steinwender C, Stuteville M, Ediebah D, Sudhir K, Bartorelli AL; ABSORB EXTEND investigators. Three-year clinical outcomes of patients treated with everolimus-eluting bioresorbable vascular scaffolds: Final results of the ABSORB EXTEND trial. Catheter Cardiovasc Interv. 2019 Jan 1;93(1):E1-E7. doi: 10.1002/ccd.27715. Epub 2018 Oct 4. PMID 30286520
- [Derived] Moriyama N, Shishido K, Tanaka Y, Yokota S, Hayashi T, Miyashita H, Koike T, Yokoyama H, Takada T, Nishimoto T, Ochiai T, Tobita K, Yamanaka F, Mizuno S, Murakami M, Takahashi S, Saito S. Neoatherosclerosis 5 Years After Bioresorbable Vascular Scaffold Implantation. J Am Coll Cardiol. 2018 May 1;71(17):1882-1893. doi: 10.1016/j.jacc.2018.02.051. PMID 29699614
- [Derived] Ishibashi Y, Nakatani S, Sotomi Y, Suwannasom P, Grundeken MJ, Garcia-Garcia HM, Bartorelli AL, Whitbourn R, Chevalier B, Abizaid A, Ormiston JA, Rapoza RJ, Veldhof S, Onuma Y, Serruys PW. Relation Between Bioresorbable Scaffold Sizing Using QCA-Dmax and Clinical Outcomes at 1 Year in 1,232 Patients From 3 Study Cohorts (ABSORB Cohort B, ABSORB EXTEND, and ABSORB II). JACC Cardiovasc Interv. 2015 Nov;8(13):1715-26. doi: 10.1016/j.jcin.2015.07.026. PMID 26585622
- [Derived] Abizaid A, Ribamar Costa J Jr, Bartorelli AL, Whitbourn R, van Geuns RJ, Chevalier B, Patel T, Seth A, Stuteville M, Dorange C, Cheong WF, Sudhir K, Serruys PW; ABSORB EXTEND investigators. The ABSORB EXTEND study: preliminary report of the twelve-month clinical outcomes in the first 512 patients enrolled. EuroIntervention. 2015 Apr;10(12):1396-401. doi: 10.4244/EIJV10I12A243. PMID 24769555
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650
- [Derived] Gogas BD, King SB 3rd, Timmins LH, Passerini T, Piccinelli M, Veneziani A, Kim S, Molony DS, Giddens DP, Serruys PW, Samady H. Biomechanical assessment of fully bioresorbable devices. JACC Cardiovasc Interv. 2013 Jul;6(7):760-1. doi: 10.1016/j.jcin.2013.04.008. No abstract available. PMID 23866188
- [Derived] Muramatsu T, Onuma Y, Garcia-Garcia HM, Farooq V, Bourantas CV, Morel MA, Li X, Veldhof S, Bartorelli A, Whitbourn R, Abizaid A, Serruys PW; ABSORB-EXTEND Investigators. Incidence and short-term clinical outcomes of small side branch occlusion after implantation of an everolimus-eluting bioresorbable vascular scaffold: an interim report of 435 patients in the ABSORB-EXTEND single-arm trial in comparison with an everolimus-eluting metallic stent in the SPIRIT first and II trials. JACC Cardiovasc Interv. 2013 Mar;6(3):247-57. doi: 10.1016/j.jcin.2012.10.013. PMID 23517836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 812 subjects (Intent-to-treat population) have been registered in 25 countries across the globe in compliance with the study Clinical Investigation Plan (CIP).
Pre-assignment Details: Out of the 812 subjects registered, a total of 43 subjects discontinued the study due to death (n=29) , withdrawal of consent (n=1) and lost-to-follow-up or missed the final 3 year follow-up visit (n=13).
Period: 30-day Follow-up Visit
Arm/Group | ABSORB BVS
Started | 812 (Intent-to-treat population (ITT).)
Completed | 812
Not Completed | 0
Period: 180-day Clinical Follow-up
Arm/Group | ABSORB BVS
Started | 812
Completed | 812
Not Completed | 0
Period: 1 - Year Visit
Arm/Group | ABSORB BVS
Started | 812
Completed | 812
Not Completed | 0
Period: 2 - Year Visit
Arm/Group | ABSORB BVS
Started | 812
Completed | 812
Not Completed | 0
Period: 3 - Year Visit
Arm/Group | ABSORB BVS
Started | 812
Completed | 769
Not Completed | 43
Not completed — Death | 29
Not completed — Withdrawal of consent | 1
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.12 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209
  Male | 603
Region of Enrollment [Number; unit: participants]
  Singapore | 20
  Malaysia | 23
  Austria | 24
  Netherlands | 67
  Sweden | 3
  Hong Kong | 21
  Brazil | 97
  Poland | 13
  France | 57
  Argentina | 20
  Japan | 40
  United Kingdom | 12
  Switzerland | 13
  India | 100
  Spain | 13
  New Zealand | 23
  Canada | 27
  Belgium | 21
  Taiwan | 74
  Denmark | 15
  Italy | 21
  South Africa | 4
  Israel | 13
  Australia | 62
  Germany | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: The composite endpoint composed of
  * Cardiac death,
  * Myocardial infarction (MI, classified as Q-wave and Non-Q wave MI),
  * Ischemia-driven target lesion revascularization (TLR) by Coronary artery bypass grafting (CABG) or Percutaneous Coronary Intervention (PCI).
Time Frame: ≤ 7 days post index procedure (In hospital)
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 14

2. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: The composite endpoint composed of
  * Cardiac death,
  * Myocardial infarction (MI, classified as Q-wave and Non-Q wave MI),
  * Ischemia-driven target lesion revascularization (TLR) by CABG or PCI.
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 21

3. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction and ischemia-driven target lesion revascularization (ID-TLR).
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 28

4. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: as for outcome 3
Time Frame: 0 to 1 year
Population: ITT population (per subject analysis). Subjects with the required follow-up are only counted once for each type of event in each time period. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 41

5. Secondary Outcome: Clinical Device Success
Description: Defined as successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis < 50% by QCA (by visual estimation if QCA is unavailable). Standard pre-dilation catheters and post-dilatation catheters (if applicable) may be used. Bailout subjects will be included as device success only if the above criteria for clinical device success are met.
Time Frame: On day 0 (immediate post-index procedure)
Population: ITT population (Per Lesion analysis). Subjects with the required follow-up are only counted once for each type of event in each time period. Subjects without the required follow-up are excluded from the time period.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Target Lesions
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 809
Number analyzed (Target Lesions) | 871
percentage of lesions | 98.9

6. Secondary Outcome: Clinical Procedure Success
Description: Defined as successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of < 50% by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of ischemia driven major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days post index procedure. In a dual lesion setting both lesions must meet clinical procedure success.
Time Frame: On day 0 (immediate post-index procedure)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 809
percentage of participants | 97.0

7. Secondary Outcome: Number of Participants With Cardiac Death
Description: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 0

8. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: Q wave MI : Development of new, pathological Q wave on the ECG Non-Q wave MI : Elevation of creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 14

9. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: Revascularization at the target lesion associated with any of the following:
  * Positive functional ischemia study.
  * Ischemic symptoms and angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA).
  * Revascularization of a target lesion with diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 0

10. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: Revascularization in the target vessel associated with any of the following:
  * Positive functional ischemia study.
  * Ischemic symptoms and an angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA).
  * Revascularization of a target vessel with diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 0

11. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 0

12. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 7
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 2

13. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: Q wave MI : Development of new, pathological Q wave on the ECG Non-Q wave MI : Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 20

14. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 4

15. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 10
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 4

16. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 0

17. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 7
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 4

18. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: as for outcome 13
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 24

19. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 9

20. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 10
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 11

21. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 4

22. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 7
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 6

23. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: as for outcome 13
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 27

24. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 19

25. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 10
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 23

26. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 10

27. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 7
Time Frame: 0 to 2 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 10

28. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: as for outcome 13
Time Frame: 0 to 2 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 35

29. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 0 to 2 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 34

30. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 10
Time Frame: 0 to 2 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 46

31. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: 0 to 2 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 20

32. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 7
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 17

33. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) - Per Protocol
Description: as for outcome 13
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
percentage of participants | 39

34. Secondary Outcome: Number of Participants With Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 9
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 41

35. Secondary Outcome: Number of Participants With Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 10
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 41

36. Secondary Outcome: Number of Participants With Ischemic Driven Non-target Lesion Target Vessel Revascularization (ID-Non-TL TVR)
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 23

37. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: The composite endpoint composed of
  * Cardiac death,
  * Myocardial infarction (Q wave and Non-Q wave),
  * Ischemia-driven target vessel revascularization by CABG or PCI.
Time Frame: ≤ 7 days post index procedure (In hospital)
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 14

38. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: as for outcome 37
Time Frame: 0 to 30 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 21

39. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: as for outcome 37
Time Frame: 0 to 180 days
Population: ITT population (per subject analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants | 30

40. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: as for outcome 37
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants | 45

41. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: as for outcome 37
Time Frame: 0 to 2 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 68

42. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF; Cardiac Death, Protocol MI, ID-TLR, ID-Non-TLR TVR)
Description: as for outcome 37
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 85

43. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: as for outcome 3
Time Frame: 0 to 2 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 807
Participants | 58

44. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE; Cardiac Death, Protocol MI, ID-TLR)
Description: as for outcome 3
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 801
Participants | 74

45. Secondary Outcome: Number of Participants With Scaffold Thrombosis (Early)
Description: According to the Academic Research Consortium (ARC) Definition, Stent Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the Catheterization lab.
  Timing:
  Acute stent thrombosis*: 0 - 24 hours post stent implantation Subacute stent thrombosis*: >24 hours - 30 days post stent implantation Late stent thrombosis†: 30 days - 1 year post stent implantation Very late stent thrombosis†: >1 year post stent implantation
  *Acute/subacute can also be replaced by early stent thrombosis. Early stent thrombosis (0 - 30 days).
  †Including "primary" as well as "secondary" late stent thrombosis; "secondary" late stent thrombosis is a stent thrombosis after a target segment revascularization.
Time Frame: 0 to 30 days
Population: ITT population (Per Subject Analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 812
Participants
  Definite | 4
  Probable | 1
  Possible | 0

46. Secondary Outcome: Number of Participants With Scaffold Thrombosis
Description: According to the ARC Definition, Stent Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the Catheterization lab.
  Timing:
  Acute stent thrombosis*: 0 - 24 hours post stent implantation Subacute stent thrombosis*: >24 hours - 30 days post stent implantation Late stent thrombosis†: 30 days - 1 year post stent implantation Very late stent thrombosis†: >1 year post stent implantation
  *Acute/subacute can also be replaced by early stent thrombosis. Early stent thrombosis (0 - 30 days).
  †Including "primary" as well as "secondary" late stent thrombosis; "secondary" late stent thrombosis is a stent thrombosis after a target segment revascularization.
Time Frame: 0 to 180 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 811
Participants
  Definite | 6
  Probable | 1
  Possible | 2

47. Secondary Outcome: Number of Participants With Scaffold Thrombosis (Late)
Description: as for outcome 46
Time Frame: 31 - 365 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 806
Participants
  Definite | 3
  Probable | 0
  Possible | 3

48. Secondary Outcome: Number of Participants With Scaffold Thrombosis
Description: as for outcome 46
Time Frame: 0 to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 808
Participants
  Definite | 7
  Probable | 1
  Possible | 3

49. Secondary Outcome: Number of Participants With Scaffold Thrombosis (Very Late)
Description: as for outcome 46
Time Frame: 366 days to 2 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 794
Participants
  Definite | 4
  Probable | 0
  Possible | 3

50. Secondary Outcome: Number of Participants With Scaffold Thrombosis
Description: as for outcome 46
Time Frame: 0 to 2 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 799
Participants
  Definite | 11
  Probable | 1
  Possible | 6

51. Secondary Outcome: Number of Participants With Scaffold Thrombosis
Description: as for outcome 46
Time Frame: 0 to 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 788
Participants
  Definite | 13
  Probable | 4
  Possible | 11

52. Secondary Outcome: Area Stenosis (%)
Time Frame: 18 months
Population: Multislice computed tomography (MSCT) subgroup. A subset of up to 100 subjects who receive at least one Absorb BVS at selected sites with MSCT capability will be assessed using MSCT at 18 months. Subjects are only counted once for each type of event in each time period.Subjects without the required follow-up are excluded from the time period.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
Percentage | 24.71 (20.55)

53. Secondary Outcome: Minimum Lumen Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 3.47 (1.04)

54. Secondary Outcome: Mean Vessel Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 13.77 (3.78)

55. Secondary Outcome: Minimum Vessel Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 9.9 (3.0)

56. Secondary Outcome: Maximum Vessel Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 18.3 (5.3)

57. Secondary Outcome: Mean Lumen Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 4.92 (1.14)

58. Secondary Outcome: Maximum Lumen Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 6.59 (1.53)

59. Secondary Outcome: Mean Plaque Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 8.85 (3.73)

60. Secondary Outcome: Minimum Plaque Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 5.41 (2.59)

61. Secondary Outcome: Maximum Plaque Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 13.18 (5.39)

62. Secondary Outcome: Mean Reference Area
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm^2 | 4.78 (1.45)

63. Secondary Outcome: Calculated Minimum Lumen Diameter
Description: The average of two orthogonal views (when possible) of the narrowest point within the area of assessment - treated lesion, treated site or treated segment. MLD is visually estimated during angiography by the Investigator; it is measured during QCA by the Angiographic Core Lab.
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
mm | 2.08 (0.32)

64. Secondary Outcome: Calculated Diameter Stenosis
Description: The value calculated as 100 * (1 - Minimum Lumen Diameter (MLD) / reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: 18 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Arm/Group | ABSORB BVS
Number analyzed (Participants) | 97
Percent Diameter stenosis | 14.05 (11.96)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | ABSORB BVS
All-Cause Mortality (participants affected / at risk) | 7/812
Serious Adverse Events (participants affected / at risk) | 295/812
Other Adverse Events (participants affected / at risk) | 808/812
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABSORB BVS (N=812)
ANEMIA (Blood and lymphatic system disorders) | 5
HEMORRHAGIC ANEMIA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANEMIA (Blood and lymphatic system disorders) | 1
NEUTROPHILIA (Blood and lymphatic system disorders) | 0
SPONTANEOUS HEMATOMA (Blood and lymphatic system disorders) | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 6
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 21
ANGINA PECTORIS (Cardiac disorders) | 80
ANGINA UNSTABLE (Cardiac disorders) | 12
ARRHYTHMIA (Cardiac disorders) | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 7
ATRIAL FLUTTER (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 3
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2
CARDIAC TAMPONADE (Cardiac disorders) | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 6
CORONARY ARTERY DISSECTION (Cardiac disorders) | 9
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2
CORONARY ARTERY STENOSIS (Cardiac disorders) | 4
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 2
INTRACARDIAC THROMBUS (Cardiac disorders) | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 7
MYOCARDIAL ISCHEMIA (Cardiac disorders) | 3
PALPITATIONS (Cardiac disorders) | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 1
PERICARDITIS (Cardiac disorders) | 1
SICK SINUS SYNDROME (Cardiac disorders) | 2
SINUS ARREST (Cardiac disorders) | 0
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0
TACHYCARDIA (Cardiac disorders) | 0
VENTRICULAR EXTRA SYSTOLES (Cardiac disorders) | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2
THYROGLOSSAL CYST (Congenital, familial and genetic disorders) | 1
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 0
TINNITUS (Ear and labyrinth disorders) | 0
VERTIGO (Ear and labyrinth disorders) | 1
GOITER (Endocrine disorders) | 1
PRIMARY HYPERALDOSTERONISM (Endocrine disorders) | 1
CATARACT (Eye disorders) | 2
CATARACT NUCLEAR (Eye disorders) | 0
DRY EYE (Eye disorders) | 0
UVEITIS (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 0
VITREOUS DEGENERATION (Eye disorders) | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0
ABDOMINAL WALL DISORDER (Gastrointestinal disorders) | 0
COLON CANCER (Gastrointestinal disorders) | 1
COLONIC POLYP (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 2
DIARRHEA (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTRIC ULCER HEMORRHAGE (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 0
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 4
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0
GINGIVITIS (Gastrointestinal disorders) | 0
GLOSSODYNIA (Gastrointestinal disorders) | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0
MELAENA (Gastrointestinal disorders) | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0
NAUSEA (Gastrointestinal disorders) | 0
PANCREATITIS (Gastrointestinal disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
TOOTH SOCKET HAEMORRHAGE (Gastrointestinal disorders) | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 4
VOMITING (Gastrointestinal disorders) | 0
ADVERSE DRUG REACTION (General disorders) | 0 — General disorders and administration site conditions
ASTHENIA (General disorders) | 1 — General disorders and administration site conditions
CATHETER SITE HAEMATOMA (General disorders) | 0 — General disorders and administration site conditions
CATHETER SITE HAEMORRHAGE (General disorders) | 0 — General disorders and administration site conditions
CATHETER SITE PAIN (General disorders) | 0 — General disorders and administration site conditions
CATHETER SITE RELATED REACTION (General disorders) | 0 — General disorders and administration site conditions
CATHETER SITE SWELLING (General disorders) | 0 — General disorders and administration site conditions
CHEST DISCOMFORT (General disorders) | 4 — General disorders and administration site conditions
CHEST PAIN (General disorders) | 5 — General disorders and administration site conditions
CHILLS (General disorders) | 0 — General disorders and administration site conditions
DEATH (General disorders) | 4 — General disorders and administration site conditions
DEVICE DISLOCATION (General disorders) | 0 — General disorders and administration site conditions
DEVICE MALFUNCTION (General disorders) | 2 — General disorders and administration site conditions
DEVICE OCCLUSION (General disorders) | 1 — General disorders and administration site conditions
DROWNING (General disorders) | 1 — General disorders and administration site conditions
FATIGUE (General disorders) | 0 — General disorders and administration site conditions
GENERAL SYMPTOM (General disorders) | 0 — General disorders and administration site conditions
MALAISE (General disorders) | 0 — General disorders and administration site conditions
MASS (General disorders) | 0 — General disorders and administration site conditions
NON-CARDIAC CHEST PAIN (General disorders) | 20 — General disorders and administration site conditions
OEDEMA (General disorders) | 0 — General disorders and administration site conditions
OEDEMA PERIPHERAL (General disorders) | 0 — General disorders and administration site conditions
PAIN (General disorders) | 0 — General disorders and administration site conditions
PYREXIA (General disorders) | 3 — General disorders and administration site conditions
SUDDEN CARDIAC DEATH (General disorders) | 2 — General disorders and administration site conditions
SUDDEN DEATH (General disorders) | 1 — General disorders and administration site conditions
THROMBOSIS IN DEVICE (General disorders) | 6 — General disorders and administration site conditions
VESSEL PUNCTURE SITE HAEMORRHAGE (General disorders) | 0 — General disorders and administration site conditions
CHOLECYSTITIS (Hepatobiliary disorders) | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 4
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0
LIVER DISORDER (Hepatobiliary disorders) | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0
HYPERSENSITIVITY (Immune system disorders) | 0
ABSCESS LIMB (Infections and infestations) | 1
BACTERIAL SEPSIS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 0
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0
DIVERTICULITIS (Infections and infestations) | 1
EMPYEMA (Infections and infestations) | 0
GASTROENTERITIS (Infections and infestations) | 3
GASTROINTESTINAL INFECTION (Infections and infestations) | 0
GROIN ABSCESS (Infections and infestations) | 0
HERPES SIMPLEX (Infections and infestations) | 0
HERPES ZOSTER (Infections and infestations) | 0
INFECTED BITES (Infections and infestations) | 0
INFLUENZA (Infections and infestations) | 0
KIDNEY INFECTION (Infections and infestations) | 0
LIVER ABSCESS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 3
LYMPHANGITIS (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 0
NOSOCOMIAL INFECTION (Infections and infestations) | 0
OSTEOMYELITIS (Infections and infestations) | 1
OSTEOMYELITIS ACUTE (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 6
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1
RASH PUSTULAR (Infections and infestations) | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
SEPSIS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 0
TUBERCULOSIS (Infections and infestations) | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0
URINARY TRACT INFECTION (Infections and infestations) | 3
VARICELLA (Infections and infestations) | 0
VIRAL INFECTION (Infections and infestations) | 0
WOUND INFECTION (Infections and infestations) | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0
BACK INJURY (Injury, poisoning and procedural complications) | 1
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0
CONTUSION (Injury, poisoning and procedural complications) | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 0
FALL (Injury, poisoning and procedural complications) | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
FOREIGN BODY (Injury, poisoning and procedural complications) | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 7
INJURY (Injury, poisoning and procedural complications) | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0
LACERATION (Injury, poisoning and procedural complications) | 1
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 10
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 0
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 0
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 0
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
TENDON INJURY (Injury, poisoning and procedural complications) | 1
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 3
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 0
BLOOD CREATININE INCREASED (Investigations) | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0
BLOOD PRESSURE ABNORMAL (Investigations) | 0
BLOOD PRESSURE DECREASED (Investigations) | 0
BLOOD PRESSURE INCREASED (Investigations) | 0
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 1
CARDIAC ENZYMES INCREASED (Investigations) | 2
CARDIAC STRESS TEST ABNORMAL (Investigations) | 3
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 0
FEMORAL BRUIT (Investigations) | 0
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 0
HEART RATE INCREASED (Investigations) | 0
HEPATIC ENZYME INCREASED (Investigations) | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 0
OXYGEN SATURATION DECREASED (Investigations) | 0
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 0
TROPONIN I INCREASED (Investigations) | 0
TROPONIN INCREASED (Investigations) | 0
TROPONIN T INCREASED (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 0
GOUT (Metabolism and nutrition disorders) | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1
JAW CYST (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
HAIR FOLLICLE TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MEDIASTINUM NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RETROPERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1
BALANCE DISORDER (Nervous system disorders) | 0
BURNING SENSATION (Nervous system disorders) | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 4
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0
CEREBRAL HAEMATOMA (Nervous system disorders) | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5
DEMENTIA (Nervous system disorders) | 0
DIZZINESS (Nervous system disorders) | 1
DIZZINESS POSTURAL (Nervous system disorders) | 0
ENCEPHALITIS (Nervous system disorders) | 1
EXERTIONAL HEADACHE (Nervous system disorders) | 0
HEADACHE (Nervous system disorders) | 0
HYPOAESTHESIA (Nervous system disorders) | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1
LETHARGY (Nervous system disorders) | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 0
PARAESTHESIA (Nervous system disorders) | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0
PARKINSONISM (Nervous system disorders) | 1
PRESYNCOPE (Nervous system disorders) | 3
SYNCOPE (Nervous system disorders) | 4
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 5
TREMOR (Nervous system disorders) | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0
DELIRIUM (Psychiatric disorders) | 0
DEPRESSION (Psychiatric disorders) | 2
INSOMNIA (Psychiatric disorders) | 0
MAJOR DEPRESSION (Psychiatric disorders) | 1
MANIA (Psychiatric disorders) | 1
MENTAL DISORDER (Psychiatric disorders) | 1
MOOD SWINGS (Psychiatric disorders) | 0
NERVOUSNESS (Psychiatric disorders) | 0
PANIC ATTACK (Psychiatric disorders) | 0
RESTLESSNESS (Psychiatric disorders) | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1
BLADDER DILATATION (Renal and urinary disorders) | 0
BLADDER OBSTRUCTION (Renal and urinary disorders) | 1
CALCULUS URINARY (Renal and urinary disorders) | 1
DYSURIA (Renal and urinary disorders) | 0
POLLAKIURIA (Renal and urinary disorders) | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2
RENAL COLIC (Renal and urinary disorders) | 2
RENAL FAILURE (Renal and urinary disorders) | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 0
RENAL MASS (Renal and urinary disorders) | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0
IDIOPATHIC URTICARIA (Skin and subcutaneous tissue disorders) | 0
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0
RASH (Skin and subcutaneous tissue disorders) | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0
OCCUPATIONAL EXPOSURE TO AIR CONTAMINANTS (Social circumstances) | 0
CARDIAC ABLATION (Surgical and medical procedures) | 1
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 1
CHOLECYSTECTOMY (Surgical and medical procedures) | 1
FLUID REPLACEMENT (Surgical and medical procedures) | 1
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 1
PROSTATECTOMY (Surgical and medical procedures) | 1
TOOTH EXTRACTION (Surgical and medical procedures) | 0
URETHRAL STENT REMOVAL (Surgical and medical procedures) | 1
VASECTOMY (Surgical and medical procedures) | 0
AORTIC ANEURYSM (Vascular disorders) | 1
BLOOD PRESSURE INADEQUATELY CONTROLLED (Vascular disorders) | 0
HAEMATOMA (Vascular disorders) | 0
HAEMORRHAGE (Vascular disorders) | 0
HYPERTENSION (Vascular disorders) | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 2
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2
PERIPHERAL COLDNESS (Vascular disorders) | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 2
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1
VENOUS INSUFFICIENCY (Vascular disorders) | 1
VENOUS THROMBOSIS (Vascular disorders) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABSORB BVS (N=812)
ANEMIA (Blood and lymphatic system disorders) | 4
HEMORRHAGIC ANEMIA (Blood and lymphatic system disorders) | 0
IRON DEFICIENCY ANEMIA (Blood and lymphatic system disorders) | 0
NEUTROPHILIA (Blood and lymphatic system disorders) | 1
SPONTANEOUS HEMATOMA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 66
ANGINA UNSTABLE (Cardiac disorders) | 4
ARRHYTHMIA (Cardiac disorders) | 3
ARTERIOSPASM CORONARY (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 9
ATRIAL FLUTTER (Cardiac disorders) | 2
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0
BRADYCARDIA (Cardiac disorders) | 5
CARDIAC ARREST (Cardiac disorders) | 0
CARDIAC FAILURE (Cardiac disorders) | 2
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0
CORONARY ARTERY DISSECTION (Cardiac disorders) | 16
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 0
INTRACARDIAC THROMBUS (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0
MYOCARDIAL ISCHEMIA (Cardiac disorders) | 0
PALPITATIONS (Cardiac disorders) | 8
PERICARDIAL EFFUSION (Cardiac disorders) | 1
PERICARDITIS (Cardiac disorders) | 0
SICK SINUS SYNDROME (Cardiac disorders) | 0
SINUS ARREST (Cardiac disorders) | 1
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 2
VENTRICULAR EXTRA SYSTOLES (Cardiac disorders) | 3
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
THYROGLOSSAL CYST (Congenital, familial and genetic disorders) | 0
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 2
GOITER (Endocrine disorders) | 1
PRIMARY HYPERALDOSTERONISM (Endocrine disorders) | 0
CATARACT (Eye disorders) | 1
CATARACT NUCLEAR (Eye disorders) | 1
DRY EYE (Eye disorders) | 2
UVEITIS (Eye disorders) | 0
VISION BLURRED (Eye disorders) | 1
VITREOUS DEGENERATION (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 4
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6
ABDOMINAL WALL DISORDER (Gastrointestinal disorders) | 1
COLON CANCER (Gastrointestinal disorders) | 0
COLONIC POLYP (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 3
DIARRHEA (Gastrointestinal disorders) | 11
DYSPEPSIA (Gastrointestinal disorders) | 5
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0
GASTRIC ULCER HEMORRHAGE (Gastrointestinal disorders) | 0
GASTRITIS (Gastrointestinal disorders) | 5
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1
GINGIVITIS (Gastrointestinal disorders) | 1
GLOSSODYNIA (Gastrointestinal disorders) | 1
HEMATOCHEZIA (Gastrointestinal disorders) | 0
HEMORRHOIDS (Gastrointestinal disorders) | 4
INGUINAL HERNIA (Gastrointestinal disorders) | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 2
MELENA (Gastrointestinal disorders) | 0
MOUTH HEMORRHAGE (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 6
PANCREATITIS (Gastrointestinal disorders) | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0
PERITONEAL HEMORRHAGE (Gastrointestinal disorders) | 0
SMALL INTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0
TOOTH SOCKET HEMORRHAGE (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0
VOMITING (Gastrointestinal disorders) | 1
ADVERSE DRUG REACTION (General disorders) | 27
ASTHENIA (General disorders) | 6 — General disorders and administration site conditions
CATHETER SITE HAEMATOMA (General disorders) | 40 — General disorders and administration site conditions
CATHETER SITE HAEMORRHAGE (General disorders) | 17 — General disorders and administration site conditions
CATHETER SITE PAIN (General disorders) | 12 — General disorders and administration site conditions
CATHETER SITE RELATED REACTION (General disorders) | 2 — General disorders and administration site conditions
CATHETER SITE SWELLING (General disorders) | 1 — General disorders and administration site conditions
CHEST DISCOMFORT (General disorders) | 13 — General disorders and administration site conditions
CHEST PAIN (General disorders) | 7 — General disorders and administration site conditions
CHILLS (General disorders) | 1 — General disorders and administration site conditions
DEVICE DISLOCATION (General disorders) | 2 — General disorders and administration site conditions
DEVICE MALFUNCTION (General disorders) | 0 — General disorders and administration site conditions
DEVICE OCCLUSION (General disorders) | 0 — General disorders and administration site conditions
DROWNING (General disorders) | 0 — General disorders and administration site conditions
FATIGUE (General disorders) | 16 — General disorders and administration site conditions
GENERAL SYMPTOM (General disorders) | 1 — General disorders and administration site conditions
MALAISE (General disorders) | 1 — General disorders and administration site conditions
MASS (General disorders) | 1 — General disorders and administration site conditions
NON-CARDIAC CHEST PAIN (General disorders) | 63 — General disorders and administration site conditions
OEDEMA (General disorders) | 1 — General disorders and administration site conditions
OEDEMA PERIPHERAL (General disorders) | 7 — General disorders and administration site conditions
PAIN (General disorders) | 1 — General disorders and administration site conditions
PYREXIA (General disorders) | 6 — General disorders and administration site conditions
THROMBOSIS IN DEVICE (General disorders) | 0 — General disorders and administration site conditions
VESSEL PUNCTURE SITE HAEMORRHAGE (General disorders) | 1 — General disorders and administration site conditions
CHOLECYSTITIS (Hepatobiliary disorders) | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
LIVER DISORDER (Hepatobiliary disorders) | 1
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 1
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 0
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 4
HYPERSENSITIVITY (Immune system disorders) | 4
ABSCESS LIMB (Infections and infestations) | 0
BACTERIAL SEPSIS (Infections and infestations) | 0
BRONCHITIS (Infections and infestations) | 3
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 0
EMPYEMA (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
GASTROINTESTINAL INFECTION (Infections and infestations) | 2
GROIN ABSCESS (Infections and infestations) | 1
HERPES SIMPLEX (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 3
INFECTED BITES (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 2
KIDNEY INFECTION (Infections and infestations) | 1
LIVER ABSCESS (Infections and infestations) | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
LUNG INFECTION (Infections and infestations) | 1
LYMPHANGITIS (Infections and infestations) | 0
NASOPHARYNGITIS (Infections and infestations) | 4
NOSOCOMIAL INFECTION (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 0
OSTEOMYELITIS ACUTE (Infections and infestations) | 0
PNEUMONIA (Infections and infestations) | 3
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0
RASH PUSTULAR (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 0
SEPTIC SHOCK (Infections and infestations) | 0
TOOTH INFECTION (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
URINARY TRACT INFECTION (Infections and infestations) | 4
VARICELLA (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
BACK INJURY (Injury, poisoning and procedural complications) | 0
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0
CATHETER SITE HAEMATOMA (Injury, poisoning and procedural complications) | 3
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 3
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0
FOREIGN BODY (Injury, poisoning and procedural complications) | 0
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 3
INJURY (Injury, poisoning and procedural complications) | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 2
LACERATION (Injury, poisoning and procedural complications) | 2
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 13
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 0
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 2
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 4
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 4
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 7
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0
TENDON INJURY (Injury, poisoning and procedural complications) | 0
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 18
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 39
BLOOD CREATININE INCREASED (Investigations) | 2
BLOOD GLUCOSE INCREASED (Investigations) | 3
BLOOD PRESSURE ABNORMAL (Investigations) | 1
BLOOD PRESSURE DECREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 3
C-REACTIVE PROTEIN INCREASED (Investigations) | 2
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 0
CARDIAC ENZYMES INCREASED (Investigations) | 50
CARDIAC STRESS TEST ABNORMAL (Investigations) | 0
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 2
FEMORAL BRUIT (Investigations) | 1
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 2
HEART RATE INCREASED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 3
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 1
OXYGEN SATURATION DECREASED (Investigations) | 2
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 1
TROPONIN I INCREASED (Investigations) | 43
TROPONIN INCREASED (Investigations) | 71
TROPONIN T INCREASED (Investigations) | 31
DIABETES MELLITUS (Metabolism and nutrition disorders) | 9
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 17
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0
JAW CYST (Musculoskeletal and connective tissue disorders) | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
HAIR FOLLICLE TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
MEDIASTINUM NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
RETROPERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0
BALANCE DISORDER (Nervous system disorders) | 1
BURNING SENSATION (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2
CEREBRAL HAEMATOMA (Nervous system disorders) | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0
DEMENTIA (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 12
DIZZINESS POSTURAL (Nervous system disorders) | 3
ENCEPHALITIS (Nervous system disorders) | 0
EXERTIONAL HEADACHE (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 18
HYPOAESTHESIA (Nervous system disorders) | 3
ISCHAEMIC STROKE (Nervous system disorders) | 0
LETHARGY (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 0
MIGRAINE (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 3
PARKINSON'S DISEASE (Nervous system disorders) | 1
PARKINSONISM (Nervous system disorders) | 0
PRESYNCOPE (Nervous system disorders) | 13
SYNCOPE (Nervous system disorders) | 6
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3
TREMOR (Nervous system disorders) | 2
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0
ANXIETY (Psychiatric disorders) | 4
CONFUSIONAL STATE (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 3
MAJOR DEPRESSION (Psychiatric disorders) | 0
MANIA (Psychiatric disorders) | 0
MENTAL DISORDER (Psychiatric disorders) | 0
MOOD SWINGS (Psychiatric disorders) | 1
NERVOUSNESS (Psychiatric disorders) | 2
PANIC ATTACK (Psychiatric disorders) | 1
RESTLESSNESS (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0
BLADDER DILATATION (Renal and urinary disorders) | 1
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0
CALCULUS URINARY (Renal and urinary disorders) | 0
DYSURIA (Renal and urinary disorders) | 2
POLLAKIURIA (Renal and urinary disorders) | 1
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0
RENAL COLIC (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
RENAL MASS (Renal and urinary disorders) | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 1
GYNAECOMASTIA (Reproductive system and breast disorders) | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 14
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 10
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0
RALES (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 3
IDIOPATHIC URTICARIA (Skin and subcutaneous tissue disorders) | 1
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 2
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 2
PSORIASIS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 8
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2
OCCUPATIONAL EXPOSURE TO AIR CONTAMINANTS (Social circumstances) | 1
CARDIAC ABLATION (Surgical and medical procedures) | 0
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 0
CHOLECYSTECTOMY (Surgical and medical procedures) | 0
FLUID REPLACEMENT (Surgical and medical procedures) | 0
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 0
PROSTATECTOMY (Surgical and medical procedures) | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 1
URETHRAL STENT REMOVAL (Surgical and medical procedures) | 0
VASECTOMY (Surgical and medical procedures) | 1
AORTIC ANEURYSM (Vascular disorders) | 0
BLOOD PRESSURE INADEQUATELY CONTROLLED (Vascular disorders) | 1
HAEMATOMA (Vascular disorders) | 3
HAEMORRHAGE (Vascular disorders) | 2
HYPERTENSION (Vascular disorders) | 18
HYPERTENSIVE CRISIS (Vascular disorders) | 3
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0
HYPOTENSION (Vascular disorders) | 17
ILIAC ARTERY OCCLUSION (Vascular disorders) | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1
PERIPHERAL COLDNESS (Vascular disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 0
VENOUS THROMBOSIS (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less